CLINICAL TRIAL: NCT03416842
Title: Home-based Exercises Using Wearable Motion Sensors for Community-dwelling Stroke Survivors With Hemiparesis
Brief Title: Home Exercise With Wearable Sensors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: 4D Motion Sports (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BRC559
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Stroke; Hemiparesis
Keywords: outpatient; wearable sensors; home exercise
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training with 4D Motion Capture Device (Experimental): Participants will be given access to a tablet-based application and non-invasive sensors that will track movements of the upper extremity and will prompt daily exercise. Participants will be encouraged to use the device daily for 30 consecutive days, up to one hour per day.
  Interventions: Device: Training with 4D Motion Capture Device

INTERVENTIONS:
Device: Training with 4D Motion Capture Device — Participants will be given access to a tablet-based application and non-invasive sensors that will track movements of the upper extremity and will prompt daily exercise. Participants will be encouraged to use the device daily for 30 consecutive days, up to one hour per day.

SUMMARY:
Repetitious motor therapy has been shown to yield the greatest improvement in motor function in those who suffer hemiplegia because of a neurological impairment. However, motor therapy remains largely clinically based due to the absence of quantitative home-based therapy technology or equipment. With the current lack of accountability, patient adherence to home exercise physical therapy programs is estimated to be as low as 35%. In response, some companies have extended the applications of their motion capture devices to be used for home-based physical therapy. However, the technologies often have not passed their initial stages of development. In contrast, a company named 4D Motion is actively working alongside the Restorative Neurology Clinic at Burke Medical Research Institute to develop a motion capture system tailored to the motor rehabilitation of hemiplegic stroke patients. This device is driven by a user's active range of motion and does not impart electrical or mechanical stimulation to the user. The device does not force the user beyond their active range of motion and does not apply resistance to motion that limits the user's capability. The 4D Motion capture system is only used to record what the patient is doing and to promote adherence to their prescribed physical therapy plan.

ELIGIBILITY:
Inclusion Criteria:

* Able to follow 1-2 step commands
* Neurological deficit leading to hemiparesis or hemiplegia with a sensorimotor deficit
* Fugl Meyer Upper Extremity Score of at least 20/66

Exclusion Criteria:

* Has a metal implant anywhere on or inside the body
* Fixed contracture or deformity of affected upper extremity
* Individuals with bilateral stroke (i.e. if both arms are affected)
* Unable to tolerate repetitious movement as determined by Likert Scale Rating greater than 5 out of 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of treatment days completed | From day 1 to day 30 of intervention
  Measure of the number of days that the participant adheres to the prescribed therapy plan (completion of 1000 movements). Goal is to have participants perform 1000 movements per day over 30 days.
Change in active range of motion of shoulder, elbow, and wrist | From day 1 to day 30 of intervention
  Maximum angular position about a joint that the participant can reach without assistance.

SECONDARY OUTCOMES:
Change in Fugl Meyer upper extremity assessment | From day 1 to day 30 of intervention
  Clinical scale that measures upper extremity impairment in stroke patients
Physical Activity Enjoyment Scale | Day 30 of intervention
  Survey of how well a participant enjoyed the study treatment.
System usability survey | Day 30 of intervention
  Survey of user-friendliness of software and device

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No